CLINICAL TRIAL: NCT00878670
Title: Prospective Clinical Trial to Assess the Efficacy and Safety of EPOGAM 1000 in Patients With Atopic Dermatitis (Explorative Pilot Study)
Brief Title: Investigation of Efficacy and Safety of EPOGAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Max Zeller Soehne AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ze 358 2008.01
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Atopic Dermatitis; Neurodermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Neurodermatitis | interventions — evening primrose oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: EPOGAM 1000 — One capsule of EPOGAM 1000 contains 932-1073 mg Oenothera seminis oleum, equivalent to 80 mg gamma-linolic acid. Children (2-12 years) take 2 capsules in the morning and evening, whereas persons over 12 years take 3 capsules in the morning and evening. The duration of the treatment is 12 weeks.
  Other Names: Oenothera seminis oleum; Evening Primrose Oil; EPOGAM

SUMMARY:
In this study it will be investigated if patients with atopic dermatitis responding to EPOGAM treatment, show a significant increase of dihomo-gamma-linolic acid in the blood.

DETAILED DESCRIPTION:
Patients with atopic dermatitis will receive EPOGAM 1000 for 12 weeks. Clinical symptoms of the disease will be assessed using the SCORAD score. Dihomo-gamma-linolic acid levels in the blood will be measured with GC-MS.

ELIGIBILITY:
Inclusion Criteria:

* atopic dermatitis since at least 2 months (criteria after Hanifin and Rajka, 1980)
* men or women aged 2 - 45 years
* women of childbearing age using contraception
* informed consent of the patient or of the parents

Exclusion Criteria:

* psychiatric disorder
* abuse of drugs or alcohol
* chronic dermatosis
* glaucoma, cataract or ocular herpes simplex
* Immune deficiency
* Immunological diseases
* clinical relevant changes in laboratory parameters
* congenital diseases
* scabies, infections with dermathophytae, HIV-associated dermatosis
* malignant diseases
* metabolic diseases
* parasites
* patients enrolled in other studies
* progredient, systemic diseases
* pregnancy and lactation
* severe internistic diseases
* organ transplantation in the medical history
* hypersensitivity against an ingredient of the study medication

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2009-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Levels of dihomo-gamma linolic acid in the blood | 0, 4 and 12 weeks after start of treatment
Efficacy of EPOGAM 1000 treatment on the symptoms of atopic dermatitis | 0, 4 and 12 weeks after start of treatment

SECONDARY OUTCOMES:
Assessment of the efficacy of EPOGAM 1000 treatment by the patient on a visual analog scale | 4 and 12 weeks after start of treatment
Assessment of the symptoms itching, sleep disorder, skin sensation, skin condition by the patient on a visual analog scale | 4 and 12 weeks after start of treatment
Willingness of the patient to further take the medication and assessment of problems related to the intake of the study drug. | 12 weeks after start of treatment
Assessment of the efficacy of EPOGAM treatment by the investigator | 4 and 12 weeks after start of treatment
Assessment of adverse events (AE) | During treatment (12 weeks)
Physical examination | 0, 4 and 12 weeks after start of treatment
Laboratory values (blood examination) | 0, 4 and 12 weeks after start of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Grendelmeier, MD, Principal Investigator — University Clinic Zurich
Locations (2):
- Switzerland (2):
  - Children Clinic, Canton Hospital Aarau, Aarau, Canton of Aargau
  - University Hospital Zurich, Zurich, Canton of Zurich

REFERENCES:
- [Background] Henz BM, Jablonska S, van de Kerkhof PC, Stingl G, Blaszczyk M, Vandervalk PG, Veenhuizen R, Muggli R, Raederstorff D. Double-blind, multicentre analysis of the efficacy of borage oil in patients with atopic eczema. Br J Dermatol. 1999 Apr;140(4):685-8. doi: 10.1046/j.1365-2133.1999.02771.x. PMID 10233322
- [Background] Yoon S, Lee J, Lee S. The therapeutic effect of evening primrose oil in atopic dermatitis patients with dry scaly skin lesions is associated with the normalization of serum gamma-interferon levels. Skin Pharmacol Appl Skin Physiol. 2002 Jan-Feb;15(1):20-5. doi: 10.1159/000049385. PMID 11803254
- [Derived] Simon D, Eng PA, Borelli S, Kagi R, Zimmermann C, Zahner C, Drewe J, Hess L, Ferrari G, Lautenschlager S, Wuthrich B, Schmid-Grendelmeier P. Gamma-linolenic acid levels correlate with clinical efficacy of evening primrose oil in patients with atopic dermatitis. Adv Ther. 2014 Feb;31(2):180-8. doi: 10.1007/s12325-014-0093-0. Epub 2014 Jan 17. PMID 24435467